CLINICAL TRIAL: NCT03332888
Title: Phase II Clinical Trial Testing the Safety of a Humanized Monoclonal Antibody Anti-CD20 in Patients With Heart Failure With Reduced Ejection Fraction
Brief Title: Safety of HMA-CD20 in Patients With HFrEF
Acronym: ICFEr-RITU2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Cardiología y Medicina Vascular Hospital Zambrano-Hellion Tec Salud (Other)
Responsible Party: Principal Investigator, David Rodriguez, MD, Instituto de Cardiología y Medicina Vascular Hospital Zambrano-Hellion Tec Salud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICFEr-RITU2
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional Group (Experimental): For this trial, HMA-CD20 will be given as an intravenous infusion of 1000 mg I.V twice in a month separating them by fourteen days starting at the baseline visit. The dose for both HMA-CD20 dosages willbe identical at the screening visit after the participant's eligibility has been established, and it will remain thesame for both infusions. The standard dose for HMA-CD20 is 1,000 mg per intravenous infusion on day 1 and day 15.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab will be studied in patients with HFrEF, and verify the patients safety.

SUMMARY:
The study is a phase II single-centered, single group, prospective clinical trial to evaluate the safety of HMA-CD20 doses among stable patients with class III/IV according to the NYHA classification with HFrEF receiving standard of care therapy. The index qualifying HFrEF must have EF < 40% based on echocardiographic or cardiac MRI techniques, heart failure class III/IV according to the NYHA classification,aged 40-60 years, being diagnosed less than 12 months before enrollment of study, following the standard heart failure treatment regimen.

ELIGIBILITY:
4.1 Inclusion criteria

1. Men and women (women not pregnant neither in lactation period) between ≥ 40 to 60 years-old.
2. Diagnosis of HFrEF and functional class III-IV.
3. EF ≤ 40% evaluated by MRI and or transthoracic echocardiography, with validity of twelve months.
4. Inadequate response to standard treatment.
5. Urgent medical attention or hospitalization due to worsening of HF or MI in the last 12 months.
6. Diagnosis of ischemic or non ischemic dilated cardiomyopathy.
7. Life expectancy of at least six months, in investigator opinion.
8. Participants should sign an (informed consent form) ICF form personally.

4.2 Exclusion criteria

1. Severe primary valvular cardiopathy or valvular prosthesis (mechanical or bio-valve).
2. History of heart transplant surgery, cardiomyoplasty, left ventricular reduction surgery, valvuloplasty, implantation of a ventricle assist device (VAD) and surgical cardiac congenital defect correction.
3. Uncontrolled atrial fibrillation (HR > 100 bpm), atrial flutter, sustained atrial fibrillation and / or significant arrhythmias such as sustained or unsustained ventricular tachychardia, bigeminy or trigeminy evidenced by Holter during the prescreening period.
4. Implantable cardioverter defibrillator (ICD) within the last three months.
5. Acute coronary syndromes that required pharmacological or mechanical reperfusion or medical treatment, within 30 days before selection.
6. Percutaneous coronary intervention within 30 days prior to selection.
7. Treatment with inotropic agents (dobutamine, milrinone, levosimendan), I.V. diuretics or vasodilators within 30 days of selection.
8. Pregnant women or breast feeding period without adequate prenatal care.
9. Untreated thyroid disease.
10. Patients with GFR <30mL/min based on the cockcroft-gualt formula
11. Rapidly progressive glomerulonephritis, seizures or psychosis, progressive neuropathy or myopathy.
12. Hemoglobin: < 8.5 mg/dL.
13. WBC count less than 5000/mm3
14. Platelets: <100,000/mm, AST or ALT >2.5 × upper limit of normal (ULN) unless related to primary disease.
15. Positive Hepatitis B or C serology (Hep B Surface antigen and Hep C antibody).
16. History of positive HIV.
17. Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer).
18. Recipients of an available attenuated vaccine within four weeks prior to randomization.
19. Previous treatment with HMA-CD20 or any immunotherapy.
20. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
21. Known active bacterial, viral, fungal (excluding fungal infections of nail beds/onychomycosis), mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease) or any major episode of infection requiring hospitalization or treatment with I.V. antibiotics within four weeks of screening, or oral antibiotics within two weeks before screening.
22. Consistent steroid administration within the past four weeks.
23. Lack of peripheral venous access.
24. Concomitant or previous malignancies, except curatively resected non-melanoma skin carcinomas or carcinoma in situ of the cervix.
25. History of psychiatric disorder that would interfere with participation in this protocol, such as depression, bipolar syndrome, schizophrenia.
26. Patients with concomitant severe COPD or emphysema.
27. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
28. Female participants without adequate method of contraception
29. Inability to comply/assist with study and follow-up procedures.

4.3 Elimination criteria

1. Progression of NYHA functional class since the initiation of the study.
2. BNP or troponin I elevation
3. New onset of pulmonary infection due to opportunistic virulent antigens (N. Jirovecci, A. Baumanni, MRSA, VRSA).
4. Any serious adverse event (SAE) indicative of fatal or nonfatal hepatitis, liver failure or its complications.
5. ALT or AST >3x normal values with a total bilirubin ≥ 2x normal value.
6. WBC count < 3000/mm3
7. Anaphylactic or life-threatening hypersensitivity reactions

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-04-16 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Rituximab Emergent Cardiovascular Adverse Events | 6 months
  The investigators analyze the safety of rituximab based on the occurrence of cardiovascular adverse events such as arrhythmia, worsening of symptoms and acute coronary syndromes.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchez-Trujillo L, Jerjes-Sanchez C, Rodriguez D, Panneflek J, Ortiz-Ledesma C, Garcia-Rivas G, Torre-Amione G. Phase II clinical trial testing the safety of a humanised monoclonal antibody anti-CD20 in patients with heart failure with reduced ejection fraction, ICFEr-RITU2: study protocol. BMJ Open. 2019 Mar 27;9(3):e022826. doi: 10.1136/bmjopen-2018-022826. PMID 30918029